CLINICAL TRIAL: NCT01758900
Title: CO2 Versus Air Insufflation for Single-balloon Enteroscopy: a Randomized, Controlled Trial
Brief Title: CO2 Versus Air Insufflation for Single-balloon Enteroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhizheng Ge (Other)
Responsible Party: Sponsor-Investigator, Zhizheng Ge, Shanghai Institute of Digestive Disease，Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: rjer2011-70k
Record Dates: First submitted 2012-12-18; First posted 2013-01-01 (Estimated); Results first posted 2016-07-14 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-10

CONDITIONS: Intubation Depth
Keywords: Single-Balloon Enteroscopy
MeSH Terms: interventions — Pneumoradiography

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Air insufflation regulator (Active Comparator): Room air will be used for insufflation as the Active Comparator arm
  Interventions: Device: Air insufflation
- CO2 insufflation regulator (Experimental): Device: CO2 insufflation regulator
  Interventions: Device: CO2 insufflation regulator

INTERVENTIONS:
Device: CO2 insufflation regulator — The CO2 insufflation regulator is Olympus UCR(Olympus Optical Co., Ltd., Tokyo, Japan). The device connect the medical gas pipe joints and CO2 cylinders, then the CO2 gas will be pumped into the delivery tube which links to the water bottle until it insufflate the bowel through the SBE.
  Arms: CO2 insufflation regulator
Device: Air insufflation — The air will be pumped into the delivery tube which links to the water bottle until it insufflate the bowel through the SBE.
  Arms: Air insufflation regulator

SUMMARY:
Small-balloon enteroscopy is a novel endoscopy system for examination of the deep small intestine.Initial reports indicated that CO2 was effective during the colonoscopy ,ERCP(endoscopic retrograde cholangiopancreatography) and DBE(double-balloon enteroscopy) examination, but it is still uncertain to the SBE(single-balloon enteroscopy) procedure.

DETAILED DESCRIPTION:
Currently, air is more frequently used to insufflate gas into the lumen to ensure the visualization of the mucosa. However, there're some limitations, for instance, significant amounts of air are usually retained in the small bowel, which will lead to the distention and the pain of the gastrointestinal tract during and after the procedure.

Carbon dioxide(CO2), comparing to the air, is rapidly absorbed from the intestine, which allows the bowel to decompress more quickly and potentially decreases intraprocedural and postprocedural pain, sedation medication requirements, procedure time, and recovery time. It is also to the benefit of deeper intubation depth so that higher total enteroscopy rate and diagnostic rate will be achieved.

Initial reports indicated that CO2 was effective during the colonoscopy ,ERCP and DBE examination, but it is still uncertain to the SBE procedure

ELIGIBILITY:
Inclusion Criteria:

* patients referred for SBE at the trial centre

Exclusion Criteria:

* Age under 18 years, over 75 years Refusal of participation GIST(gastrointestinal stromal tumor), apparent tumor, post surgery Crohn's disease, Intestinal obstruction, stenosis, radiation enteritis Severe cardiopulmonary dysfunction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhizheng Ge, Ph.D. MD., Principal Investigator — Department of Gastroenterology, Renji Hospital, Shanghai Institute of Digestive Diseases, Shanghai Jiao Tong University School of Medicine Shanghai
Locations (1):
- Department of Gastroenterology, Renji Hospital, Shanghai Institute of Digestive Diseases, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsujikawa T, Saitoh Y, Andoh A, Imaeda H, Hata K, Minematsu H, Senoh K, Hayafuji K, Ogawa A, Nakahara T, Sasaki M, Fujiyama Y. Novel single-balloon enteroscopy for diagnosis and treatment of the small intestine: preliminary experiences. Endoscopy. 2008 Jan;40(1):11-5. doi: 10.1055/s-2007-966976. Epub 2007 Dec 4. PMID 18058613
- [Background] Kawamura T, Yasuda K, Tanaka K, Uno K, Ueda M, Sanada K, Nakajima M. Clinical evaluation of a newly developed single-balloon enteroscope. Gastrointest Endosc. 2008 Dec;68(6):1112-6. doi: 10.1016/j.gie.2008.03.1063. Epub 2008 Jul 2. PMID 18599052
- [Background] Frantz DJ, Dellon ES, Grimm IS, Morgan DR. Single-balloon enteroscopy: results from an initial experience at a U.S. tertiary-care center. Gastrointest Endosc. 2010 Aug;72(2):422-6. doi: 10.1016/j.gie.2010.03.1117. Epub 2010 Jun 11. PMID 20541189
- [Background] Domagk D, Bretthauer M, Lenz P, Aabakken L, Ullerich H, Maaser C, Domschke W, Kucharzik T. Carbon dioxide insufflation improves intubation depth in double-balloon enteroscopy: a randomized, controlled, double-blind trial. Endoscopy. 2007 Dec;39(12):1064-7. doi: 10.1055/s-2007-966990. PMID 18072057
- [Background] Dellon ES, Hawk JS, Grimm IS, Shaheen NJ. The use of carbon dioxide for insufflation during GI endoscopy: a systematic review. Gastrointest Endosc. 2009 Apr;69(4):843-9. doi: 10.1016/j.gie.2008.05.067. Epub 2009 Jan 18. PMID 19152906
- [Background] Hirai F, Beppu T, Nishimura T, Takatsu N, Ashizuka S, Seki T, Hisabe T, Nagahama T, Yao K, Matsui T, Beppu T, Nakashima R, Inada N, Tajiri E, Mitsuru H, Shigematsu H. Carbon dioxide insufflation compared with air insufflation in double-balloon enteroscopy: a prospective, randomized, double-blind trial. Gastrointest Endosc. 2011 Apr;73(4):743-9. doi: 10.1016/j.gie.2010.10.003. Epub 2011 Jan 14. PMID 21237455
- [Background] May A, Farber M, Aschmoneit I, Pohl J, Manner H, Lotterer E, Moschler O, Kunz J, Gossner L, Monkemuller K, Ell C. Prospective multicenter trial comparing push-and-pull enteroscopy with the single- and double-balloon techniques in patients with small-bowel disorders. Am J Gastroenterol. 2010 Mar;105(3):575-81. doi: 10.1038/ajg.2009.712. Epub 2010 Jan 5. PMID 20051942
- [Background] Iddan G, Meron G, Glukhovsky A, Swain P. Wireless capsule endoscopy. Nature. 2000 May 25;405(6785):417. doi: 10.1038/35013140. No abstract available. PMID 10839527
- [Background] Yamamoto H, Sekine Y, Sato Y, Higashizawa T, Miyata T, Iino S, Ido K, Sugano K. Total enteroscopy with a nonsurgical steerable double-balloon method. Gastrointest Endosc. 2001 Feb;53(2):216-20. doi: 10.1067/mge.2001.112181. PMID 11174299
- [Background] Ramchandani M, Reddy DN, Gupta R, Lakhtakia S, Tandan M, Rao GV, Darisetty S. Diagnostic yield and therapeutic impact of single-balloon enteroscopy: series of 106 cases. J Gastroenterol Hepatol. 2009 Oct;24(10):1631-8. doi: 10.1111/j.1440-1746.2009.05936.x. Epub 2009 Aug 3. PMID 19686408
- [Background] Aktas H, de Ridder L, Haringsma J, Kuipers EJ, Mensink PB. Complications of single-balloon enteroscopy: a prospective evaluation of 166 procedures. Endoscopy. 2010 May;42(5):365-8. doi: 10.1055/s-0029-1243931. Epub 2010 Feb 22. PMID 20178072
- [Background] Upchurch BR, Sanaka MR, Lopez AR, Vargo JJ. The clinical utility of single-balloon enteroscopy: a single-center experience of 172 procedures. Gastrointest Endosc. 2010 Jun;71(7):1218-23. doi: 10.1016/j.gie.2010.01.012. Epub 2010 Apr 20. PMID 20409544
- [Derived] Li X, Zhao YJ, Dai J, Li XB, Xue HB, Zhang Y, Xiong GS, Ohtsuka K, Gao YJ, Liu Q, Song Y, Fang JY, Ge ZZ. Carbon dioxide insufflation improves the intubation depth and total enteroscopy rate in single-balloon enteroscopy: a randomised, controlled, double-blind trial. Gut. 2014 Oct;63(10):1560-5. doi: 10.1136/gutjnl-2013-306069. Epub 2014 Mar 13. PMID 24626435

RESULTS

PARTICIPANT FLOW:
Groups:
- CO2(Carbon Dioxide) Insufflation Regulator: Device: CO2 insufflation regulator
  CO2 insufflation regulator: The CO2 insufflation regulator is Olympus UCR(Olympus Optical Co., Ltd., Tokyo, Japan). The device connect the medical gas pipe joints and CO2 cylinders, then the CO2 gas will be pumped into the delivery tube which links to the water bottle until it insufflate the bowel through the SBE(single-balloon enteroscopy).
Period: Overall Study
Arm/Group | CO2(Carbon Dioxide) Insufflation Regulator | Air Insufflation Regulator
Started | 106 | 108
Completed | 99 | 100
Not Completed | 7 | 8
Not completed — difficulty for further intubation | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CO2 Insufflation Regulator | Air Insufflation Regulator | Total
Number analyzed (Participants) | 106 | 108 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (14.3) | 40.5 (17.6) | 40.8 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 48 | 89
  Male | 65 | 60 | 125
Course of disease (month) [Mean (Standard Deviation); unit: months] | 13.1 (20.2) | 13.9 (22.1) | 13.5 (21.1)
indications [Number; unit: participants]
  abdominal pain | 41 | 47 | 88
  occult gastrointestinal bleeding | 41 | 38 | 79
  Diarrhoea | 11 | 14 | 25
  Abdominal distension | 7 | 5 | 12
  Weight loss | 2 | 2 | 4
  Nausea | 2 | 0 | 2
  Vomiting | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Intubation Depth
Time Frame: Within 5 minutes after the examination
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | CO2 Insufflation Regulator | Air Insufflation Regulator
Number analyzed (Participants) | 106 | 108
cm | 323.8 (64.2) | 238.3 (68.6)

2. Secondary Outcome: Total Enteroscopy Rate
Time Frame: Within 1 week after all the examinations are finished
Measure: Number; unit: participants
Arm/Group | CO2 Insufflation Regulator | Air Insufflation Regulator
Number analyzed (Participants) | 106 | 108
participants | 37 | 19

3. Secondary Outcome: Diagnostic Rate
Time Frame: Within 1 week after all the examinations are finished
Measure: Number; unit: Percentage of Participants
Arm/Group | CO2 Insufflation Regulator | Air Insufflation Regulator
Number analyzed (Participants) | 106 | 108
Percentage of Participants | 58.5 | 47.2

4. Secondary Outcome: Patient's Acceptability
Description: Acceptability was recorded on a questionnaire given to patients after the examination. Patients assessed the degree of abdominal pain/distention along a 10-cm line of the VAS(visual analogue scale), with the 0-cm point labeled "no pain/distention" on left end and the 10-cm point labeled "very severe pain/distention that cannot be tolerated" on the right end. Patients were asked to score the severity of pain/distention experienced at 1, 2, 3 and 6 hours after the completion of the entire examination.
Time Frame: 6 hours after the examination
Measure: Number; unit: participants
Arm/Group | CO2 Insufflation Regulator | Air Insufflation Regulator
Number analyzed (Participants) | 106 | 108
participants | 105 | 107

5. Secondary Outcome: Procedure Time
Time Frame: Within 5 minutes after the examination
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | CO2 Insufflation Regulator | Air Insufflation Regulator
Number analyzed (Participants) | 106 | 108
minutes
  Oral intubation | 77.9 (36.3) | 72.9 (29.9)
  Anal intubation | 86.4 (43.7) | 75.8 (30.1)
  Total enteroscopy examinations | 166.5 (69.6) | 155.1 (57.1)

6. Secondary Outcome: Abdominal Circumference
Description: To measure abdominal circumference, a tape was placed horizontally around the abdomen at the level of the middle location between the level of anterior superior iliac spine and the lower edge of costal arch, and the measurement was made at the end of a normal expiration before and after the procedure.
Time Frame: 10 minutes before/after the examination
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | CO2 Insufflation Regulator | Air Insufflation Regulator
Number analyzed (Participants) | 99 | 100
centimeter
  Before the procedure | 73.4 (9.6) | 70.3 (4.6)
  After the procedure | 74.1 (9.7) | 73.6 (3.5)

7. Secondary Outcome: Complication Rate
Time Frame: Within 1 week after all the examinations are finished
Measure: Number; unit: participants
Arm/Group | CO2 Insufflation Regulator | Air Insufflation Regulator
Number analyzed (Participants) | 106 | 108
participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse event was defined as any event that changed the health status of a patient, occurring within 30 days after enteroscopy examination.
Arm/Group | CO2 Insufflation Regulator | Air Insufflation Regulator
Serious Adverse Events (participants affected / at risk) | 1/106 | 1/108
Other Adverse Events (participants affected / at risk) | 0/106 | 0/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CO2 Insufflation Regulator (N=106) | Air Insufflation Regulator (N=108)
acute haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
acute pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No